CLINICAL TRIAL: NCT03720145
Title: Lifestyle Medicine for Depression: A Pilot Randomized Controlled Trial
Brief Title: Lifestyle Medicine for Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other); The University of Hong Kong (Other); University of Western Sydney (Other); University of Melbourne (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY003
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Depression
Keywords: Depression; Lifestyle Medicine
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): lifestyle medicine group
  Interventions: Behavioral: Lifestyle Medicine
- CAU group (No Intervention): Care-As-Usual group

INTERVENTIONS:
Behavioral: Lifestyle Medicine — Lifestyle intervention including diet, sleep, exercise, relaxation and mindfulness
  Arms: Treatment Group

SUMMARY:
This study will examine the feasibility and efficacy of lifestyle medicine for the management of depression in Chinese adult population. The main components of lifestyle intervention typically include physical activity, diet, relaxation/mindfulness, and sleep. While lifestyle medicine has been recognized for centuries as a means to improve physical health, the field of lifestyle medicine in the context of mental health is still in its infancy. In the existing literature, there is increasing evidence demonstrating the efficacy of individual components of lifestyle medicine (e.g, physical activities and sleep) on depression. However, there is very limited research on the effectiveness of an integration of multiple lifestyle adjustments on depression.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents aged ≥ 18 years;
2. Cantonese language fluency;
3. Patient Health Questionnaire (PHQ-9) score ≥ 10; and
4. Willingness to provide informed consent and comply with the trial protocol.

Exclusion Criteria:

1. Pregnancy;
2. Have suicidal ideation based on Beck Depression inventory (BDI-II) Item 9 score ≥ 2 (referral information to professional services will be provided to those who endorsed items on suicidal ideation);
3. Using medication or psychotherapy for depression;
4. Having unsafe conditions and are not recommended for exercising or a change in diet by physicians; and
5. Have major psychiatric, medical or neurocognitive disorders that make participation infeasible or interfere with the adherence to the lifestyle modification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Patient Health Questionnaire (PHQ-9) | Baseline, 1-week post-treatment and 12-week post treatment
  The PHQ-9, a 20-item questionnaire used for screening, diagnosing, monitoring and measuring the severity of depression, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day).

SECONDARY OUTCOMES:
Change in Insomnia Severity Index (ISI) | Baseline, 1-week post-treatment and 12-week post treatment
  ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.
Change in Short form Health Survey - 36 items (SF-36) | Baseline, 1-week post-treatment and 12-week post treatment
  SF-36 is used to assess the patients' general health and quality of life. It contains 36 items, measuring 8 aspects of health domains: physical functioning, social functioning, physical role limitations, emotional role limitations, mental health, vitality, bodily pain, and general health perception.
Change in Multidimensional Fatigue Inventory (MFI) | Baseline, 1-week post-treatment and 12-week post treatment
  MFI is a 20-item self-report instrument designed to measure fatigue. Ratings on a 5-point Likert scale are obtained on the dimensions of general fatigue, physical fatigue, mental fatigue, reduced motivation and reduced activity.
Change in Sheehan Disability Scale (SDS) | Baseline, 1-week post-treatment and 12-week post treatment
  SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life
Change in Depression Anxiety Stress Scales (DASS-21) | Baseline, 1-week post-treatment and 12-week post treatment
  DASS-21 is a 21-items scales, comprises three sub-scales which measures the negative emotional states of depression, anxiety, and stress, over the past week. The DASS is based on a dimensional rather than a categorical conception of psychological disorder, thus it has no direct implications for the allocation of patients to discrete diagnostic categories. However, recommended cutoffs for conventional severity labels (normal, moderate, severe) are given in the DASS Manual.

OTHER OUTCOMES:
Change in Credibility-Expectancy Questionnaire (CEQ) | Baseline and 1-week post-treatment
  The 6-item CEQ yielded ratings of treatment credibility, acceptability/satisfaction, and expectations for success.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong